CLINICAL TRIAL: NCT01958684
Title: A Non-interventional Study to Observe the Bleeding Pattern of LNG-IUS Inserted Immediately After Surgical Abortion Compared With Copper IUD
Brief Title: Bleeding Pattern Difference Between Levonorgestrel Intrauterine System (LNG-IUS) and Copper Intrauterine Devices (IUDs) Immediately Inserted After Abortion
Acronym: POST
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16954; MA1310CN (Other: company internal)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Contraception
Keywords: Bleeding pattern; LNG-IUS; Cu-IUD; postabortion
MeSH Terms: interventions — Levonorgestrel; Intrauterine Devices, Copper

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: The MIRENA intrauterine delivery system (initial release rate: 20 μg LNG /24 h)
  Interventions: Drug: Levonorgestrel IUS (Mirena, BAY86-5028)
- Group 2: Copper IUDs with different shape and with or without drugs
  Interventions: Device: Copper-IUD

INTERVENTIONS:
Drug: Levonorgestrel IUS (Mirena, BAY86-5028) — LNG-IUS once inserted will be effective for 5 years.
  Other Names: Mirena Group
  Groups: Group 1
Device: Copper-IUD — Copper-IUD once inserted will be effective for more than 10 years.
  Other Names: Cu-IUD Group
  Groups: Group 2

SUMMARY:
To observe the bleeding patterns of post-abortion immediate insertion of IUS compared to Cu-IUD over the first 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive women in good general health and requesting long-term contraception
* Applied the Cu-IUD or LNG-IUS immediately after first trimester surgical abortion
* History of regular cyclic menstrual periods
* Written ICF was obtained

Exclusion Criteria:

* Suspected septic abortion and incomplete abortion, as well as missed abortion
* The contraindications and warnings of the respective Summary of Product Characteristics of Mirena or prescribing information of Cu-IUDs must be followed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects should go through the surgical abortion should meet both inclusion and exclusion criteria. And they are willing to sign an informed consent. And all recruitment should be conducted after the decision of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The number of bleeding/spotting days assessed over the second 90-day reference period after induced abortion | Months 4 to 6
  The 90-day reference period is recommended by the WHO. Day 1 is defined as the insertion day.

SECONDARY OUTCOMES:
Menstrual bleeding intensity | up to 6 months
  It will be captured by patient dairy and measured by subjective scale as below.
  * No bleeding
  * Light bleeding
  * Normal bleeding
  * Heavy bleeding
  * Very heavy bleeding
Abortion related bleeding days | up to 1 month
Time to the first menstrual bleeding following abortion | up to 2 months
  This data will be calculated by days
Participants continuation rates of Mirena and Cu-IUD | up to 6 months
Reasons for discontinuation of Mirena and Cu-IUD | Up to 6 months
  It will be calculated by percentage
Participants satisfaction rates of Mirena and Cu-IUD | Up to 6 months
  It will be captured by satisfaction scale as below.
  * Very satisfied
  * Rather satisfied
  * neither satisfied nor dissatisfied
  * Rather unsatisfied
  * Very unsatisfied
Percentage of participants with adverse events | Up to 6 months
  Adverse events included: Pelvic inflammatory disease, Expulsion and Others.)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China

REFERENCES:
- [Derived] Chen X, Li Q, Wang X, Chen J, Lv W, Shi B, Wang H, Luo J, Li J. Bleeding pattern difference between levonorgestrel intrauterine system and copper intrauterine devices inserted immediately post-abortion: a multicenter, prospective, observational cohort study in Chinese women. Curr Med Res Opin. 2018 May;34(5):873-880. doi: 10.1080/03007995.2017.1421919. Epub 2018 Feb 7. PMID 29298525